CLINICAL TRIAL: NCT01539798
Title: Changes in Body Composition, Hematological Parameters, and Serum Biochemistry and After Rapid Intravenous Infusion or Oral Intake of 2L of 0.9% Saline Solution in Young Healthy Volunteers. A Randomized Cross-over Study
Brief Title: Body Composition and Serum Biochemistry After Intravenous Infusion or Oral Intake of Saline in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Mato Grosso (Other)
Responsible Party: Principal Investigator, Jose Eduardo de Aguilar-Nascimento, Full Professor, Federal University of Mato Grosso
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: valente_crossover; Oral versus iv saline solution (Other Grant/Funding Number: FAPEMAT- Fundação de Amparo a Pesquisa de Mato Grosso)
Record Dates: First submitted 2012-02-18; First posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Edema; Perioperative/Postoperative Complications
Keywords: Saline solution; Sodium Chloride; Hypoalbuminemia; Weight Gain
MeSH Terms: conditions — Edema; Postoperative Complications; Hypoalbuminemia; Weight Gain | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Saline (Experimental): Ingestion of 0.9% saline solution
  Interventions: Other: Oral saline
- Intravenous Saline (Active Comparator): Intravenous infusion of 0.9% saline solution
  Interventions: Other: Intravenous saline

INTERVENTIONS:
Other: Oral saline — Ingestion of 2 L of 0.9% saline solution over 1h
  Other Names: Sodium chloride solution
  Arms: Oral Saline
Other: Intravenous saline — Infusion of 2L of 0.9% saline solution over 1h
  Other Names: Sodium chloride solution
  Arms: Intravenous Saline

SUMMARY:
The investigators conducted a cross-over study to compare the response of healthy young volunteers to a rapid oral intake or intravenous infusion of 0.9% saline solution on the body composition, serum electrolytes, albumin, and hematological parameters.

The investigators hypothesized that these parameters will differently adapt depending on the route of infusion

DETAILED DESCRIPTION:
This was a cross over study including ten healthy young males (18-26 years old) with no acute or chronic illness for the last 3 months previously. They were not using any either medications or illicit drugs. Based on their body mass index (BMI) they were neither considered obese nor malnourished (BMI ranged from 22 to 27 kg/m2). They underwent the study after giving written informed consent. The study was approved by the Committee of Ethics in Research of the Julio Muller Hospital (862/CEP-HUJM/2010; Federal University of Mato Grosso, Cuiaba, Brazil). In two separate moments, all participants received in random order 2L of 0.9% saline by either the forearm vein or oral intake as follows.

Procedures The ten volunteers were fasted from midnight and they reported to the laboratory by 8-9 AM for the procedures. After having voided the bladder they were weighted to the nearest 0.1 kg and their heights were measured to the nearest 0.01 m with a estadiometer. Body mass was then calculated. Bioelectrical impedance analysis was performed with single-frequency (50 kHz) device (Bodystat 1500; Bodystat Ltd., Isle of Man, U.K.) using tetrapolar distal limb electrodes. TBW, fatty mass and lean body mass were calculated using regression equations programmed into the devices.

Firstly, a 12 gauge cannula was inserted the forearm and blood samples were collected for laboratory assays: hematocrit, hemoglobin, blood glucose, serum electrolytes (sodium, potassium, chloride and bicarbonate), albumin, creatinine, and osmolality. The volume of the urine output until 2h after the experiment was collected and measured.

Two liters of 0.9% saline were then infused over 1 hour into one of the forearm veins in all participants in supine position. An experienced anesthetist conducted the entire procedure at the laboratory. Blood pressure and pulse rate were taken every 30 minutes for 2h and the volunteers were not allowed to eat or drink during this period. After the infusion of the saline solution they were sent to void the bladder, were weighted again, and another blood sample was taken for the same assays. Another bioelectrical impedance analysis was carried out by the same manner. Two hours after the finish of the infusion they were asked to void the bladder again and the urinary output was registered.

The same volume of saline associated with a non-caloric flavor powder (Tang, Sao Paulo, Brazil) was orally ingested by the same volunteers 4 weeks after the first experiment, in the same room and following the same preparation as described. The blood samples were sent to the laboratory with a code that was broken in the end of the experiment and the data was put in a datasheet for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young males (18-26 years) bearing no acute or chronic illness for the last 3 months previously to the experiment

Exclusion Criteria:

* Use of any drugs, tobacco, alcohol 2 months prior to the experiment. The investigators also planned to exclude those who for any reason do not comply with the protocols

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Body Composition | 2 hours
  . After having voided the bladder they were weighted to the nearest 0.1 kg and their heights were measured to the nearest 0.01 m with a estadiometer. Body mass was then calculated. Bioelectrical impedance analysis was performed with single-frequency (50 kHz) device (Bodystat 1500; Bodystat Ltd., Isle of Man, U.K.) using tetrapolar distal limb electrodes. TBW, fatty mass and lean body mass were calculated using regression equations programmed into the devices

SECONDARY OUTCOMES:
Serum electrolytes | 2 hours
  Blood samples were collected before infusion and 1h after for laboratory assays: hematocrit, hemoglobin, blood glucose, serum electrolytes (sodium, potassium, chloride and bicarbonate), albumin, creatinine, and osmolality.

CONTACTS AND LOCATIONS:
Overall Officials: Jose E Aguilar-Nascimento, MD, PhD, Principal Investigator — Federal University of Mato Grosso
Locations (1):
- Hospital Universitario Julio Mullar, Cuiabá, Mato Grosso, Brazil